CLINICAL TRIAL: NCT02129699
Title: A Randomised, Open-label Phase III Trial Evaluating the Addition of Denosumab to Standard First-line Anticancer Treatment in Advanced NSCLC
Brief Title: Survival imProvement in Lung cancEr iNduced by DenOsUmab theRapy
Acronym: SPLENDOUR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Completion of recruitment was not feasible as accrual was slower than anticipated. Even if a benefit for denosumab could be shown, these results would be of very limited clinical impact by the time they would be available
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 5-12 / EORTC 08111; 2013-003156-21 (EudraCT Number); 20080166 (Other Grant/Funding Number: AMGEN); SNCTP000000954 (Registry Identifier: Swiss National Clinical Trials Portal (SNCTP))
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Results first posted 2024-04-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer Non-small Cell Stage IV
Keywords: NSCLC; stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- None, standard chemotherapy only (Other): 4 - 6 cycles of standard chemotherapy + best supportive care including any bone protective agent except denosumab.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  Interventions: Other: None, standard chemotherapy only
- Standard chemotherapy + Denosumab (Experimental): 4 - 6 cycles of standard chemotherapy + denosumab 120 mg, administered subcutaneously every 3-4 weeks until unacceptable toxicity, patient refusal, or patient's death. Denosumab should be administered on day 1 of each cycle, before or after the administration of chemotherapy. After stop of first-line chemotherapy, denosumab must be continued life-long, regardless of tumour progression and concomitantly with subsequent lines of systemic treatment, as long as tolerable for the patient.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Denosumab: 120 mg, s.c. every 3-4 weeks (in cycle 1 additional dose on day 8) until unacceptable toxicity, patient refusal or patient's death (max. 4 years 3 months).
  Other Names: XGEVA
  Arms: Standard chemotherapy + Denosumab
Other: None, standard chemotherapy only — Possible standard chemotherapies (3 weeks cycles, duration: 4 - 6 cycles):
  Cisplatin 75 mg/m2 as an infusion on day 1 Gemcitabine 1250 mg/m2 as an infusion days 1 and 8 or Carboplatin AUC 5 as an infusion on day 1 Gemcitabine 1000 mg/m2 as an infusion days 1 and 8 or Cisplatin 75 mg/m2 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1 or Carboplatin AUC 5 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1
  Arms: None, standard chemotherapy only

SUMMARY:
The purpose of this study is to investigate how well the standard treatment (platinum-based doublet chemotherapy) in combination with denosumab works compared with the standard treatment alone in patients with a type of lung cancer called "non small cell lung cancer" (NSCLC) that has spread to other parts of the body.

DETAILED DESCRIPTION:
The investigational medicinal product denosumab is a protein (monoclonal antibody) that works to slow down bone destruction caused by cancer spreading to the bone (bone metastasis). Denosumab is used in adults with cancer to prevent serious complications caused by bone metastasis (e.g., fracture, pressure on the spinal cord or the need to receive radiation therapy or surgery). Results from one study in lung cancer patients with bone metastasis suggested that adding denosumab to the standard chemotherapy may lead to a possible survival benefit.

All patients will receive standard chemotherapy consisting of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed, depending on the nature of the lung cancer, every 3 weeks for about 3-4 months:

Patients will be assigned to one of two groups, known as 'arms'.

The treatment for each arm will be as follows:

Arm A: 4 - 6 cycles of chemotherapy and best supportive care (including any bone protective agent except denosumab)

Arm B: 4 - 6 cycles of chemotherapy + denosumab 120 mg, administered subcutaneously every 3-4 weeks until unacceptable toxicity, patient refusal or patient's death. After stop of first-line chemotherapy, denosumab must be continued every 3-4 weeks lifelong, regardless of tumour progression and concomitantly with subsequent lines of systemic treatment, as long as tolerable for the patient.

Beyond primary analysis, all subjects randomised to ARM B and still benefitting from the drug will be offered denosumab at a dose of 120 mg s.c. until patient or physician elect to discontinue denosumab for any reason, and for a maximum of 2 years after the required number of events for the final analysis has been reached.

A total of 1000 patients from centers in Europe, Switzerland and Israel are expected to be enrolled in this study over a period of 37 months. The study will take approximately 56 months to be completed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced stage IV non-small cell lung carcinoma (NSCLC), according to 7th TNM classification
* Age ≥ 18 years
* ECOG performance status 0-2
* Measurable or evaluable disease (according to RECIST 1.1 criteria) assessed within 28 days from randomization.
* Availability of tumour tissue (as assessed by the local pathologist) for translational research:
* preferred: FFPE block from primary tumour or metastasis,
* alternatively: cell block
* if no block available: 10 freshly cut unstained slides.
* Adequate haematological function: neutrophils ≥ 1.5 ×109/L, platelets

  ≥ 100×109/L, and hemoglobin ≥ 9 g/dL
* Adequate liver function:
* ALT ≤ 3 × ULN ( ≤ 5 × ULN if liver metastasis are present)
* Total bilirubin < 2 x ULN
* Adequate renal function: calculated renal creatinine clearance (CrCl) ≥ 30 mL/min (according to the formula of Cockroft-Gault)
* Life expectancy of at least 3 months
* Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 7 days before enrollment. Pregnancy test has to be repeated within 14 days before treatment start.
* All sexually active men and women of childbearing potential must use an effective contraceptive method during the study treatment and for a period of at least 6 months following the last administration of trial treatment
* Written Informed Consent must be signed and dated by the patient and the investigator prior to any trial-related intervention for

  1. Trial treatment
  2. Submission of biomaterial for central testing

Exclusion Criteria:

* Patients with presence of documented sensitizing EGFR activating mutation or ALK rearrangements (screening following local standards is optional, but strongly encouraged in non-squamous histology)
* Patients with documented brain metastases (systematic screening of patients not mandatory; however, if the patient is symptomatic, brain metastases screening is recommended).
* Prior chemotherapy or molecular targeted therapy for metastatic disease.

Exceptions:

* Neoadjuvant or adjuvant chemotherapy or radio-chemotherapy are allowed if terminated more than 6 months before registration.
* Previous radical radiotherapy without systemic treatment is allowed.
* One previous line of systemic immunotherapy by checkpoint inhibitors is allowed and needs to be documented
* Concomitant treatment with immune checkpoint inhibitors
* Any investigational agent(s) within 30 days prior to randomisation
* Concurrent bisphosphonate administration
* Oral/ dental conditions (by visual inspection):
* Prior history or current evidence of osteomyelitis / osteonecrosis of the jaw
* Active dental or jaw condition which requires oral surgery
* Planned invasive dental procedure for the course of the trial
* Non-healed dental or oral surgery
* Evidence of any medical condition which would impair the ability of the patient to participate in the trial or might preclude therapy with trial drugs (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease, active infection, uncontrolled diabetes mellitus; uncontrolled arterial hypertension ≥ 160/100 mmHg, history of myocardial infarction in the last 3 months)
* Documented active infection with Hepatitis B virus or Hepatitis C virus, known infection with human immunodeficiency virus (HIV)
* Known hypersensitivity to any of the components of the treatment
* Severe, uncorrected hypocalcaemia or hypercalcaemia:
* hypercalcaemia: total calcium >3.1 mmol/l or corrected calcium (with albumin level) >3 mmol/l
* hypocalcaemia: total calcium <2 mmol/l or corrected calcium (with albumin level) < 1.9 mmol/l
* Legal incapacity or limited legal capacity
* Medical or psychological condition, including uncontrolled arterial hypertension (>160/110) despite adequate medication which in the opinion of the investigator would not permit the patient to complete the trial or sign meaningful informed consent
* Women who are pregnant or breastfeeding
* Any concurrent malignancy other than adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, in situ breast carcinoma, or prostate cancer Gleason score < 6. (Patients with a previous malignancy but without evidence of disease for ≥ 2 years will be allowed to enter the trial)
* Any previous exposure to denosumab, with the exception of a maximum of 2 previous doses of denosumab (Prolia®) more than 6 month before enrolment for osteoporosis treatment/prevention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solange Peters, MD, PhD, Study Chair — Trial Chair, CHUV Lausanne, Switzerland; Mary O'Brien, MD, Study Chair — EORTC Trial Co-Chair, Royal Marden Hospital, Sutton, UK; Sarah Danson, PhD, Study Chair — EORTC Trial Co-Chair, University of Sheffield, Sheffield, UK; Rolf Stahel, MD, Study Chair — Trial Co-Chair, University Hospital of Zuerich, Switzerland
Locations (66):
- Austria (5):
  - Univ. Klinik für Innere Medizin V, Innsbruck
  - KH der Elisabethinen Linz, Linz
  - AKH Wien, Vienna
  - Otto-Wagner-Spital Department 1, Vienna
  - Otto-Wagner-Spital Department 2, Vienna
- Belgium (4):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - University Hosptial Ghent, Ghent
  - Centre Hospitalier Regional De La Citadelle, Liège
  - Clinique et Maternite Sainte Elisabeth, Namur
- France (17):
  - Centre hospitalier universitaire d'Angers, Angers
  - Centre Hospitalier Annecy, Annecy
  - Centre Hospitalier De Beauvais, Beauvais
  - Hôpitale de la Cavale Blanche - CHRU de BREST, Brest
  - GHPSO (Sie de Creil), Creil
  - Centre Hospitalier Intercommunal Creteil, Créteil
  - Hospital Center Le Mans, Le Mans
  - Hôpital du Cluzeau, Limoges
  - CHBS Lorient, Lorient
  - Hôpital Louis Pradel, Lyon
  - Assistance Publique-Hôitaux de Marseille, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - Centre Hospitalier Universitaire Rennes, Rennes
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - CHICAS, Sisteron
  - Hôpital de Villefranche-sur-Saône, Villefranche-sur-Saône
- Germany (2):
  - ASKLEPIOS - Fachkliniken München - Gauting, München
  - Pius Hospital, Oldenburg
- Ireland (9):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Miscordia University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St James's Hospital, Dublin
  - The Adelaide and Meath Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
  - Hospital Waterford, Waterford
- Italy (4):
  - S.G Moscati Hospital, Aversa
  - IRCCS Azienda Ospedaliera Universitaria San Martino, Genova
  - San Paolo Hospital, Milan
  - Ospedale San Gerardo, Monza
- Maria Sklodowska-Curie Memorial Car, Gliwice, Poland
- Slovenia (2):
  - University Clinic Golnik, Golnik
  - Institute of Oncology Ljubljana, Ljubljana
- Spain (12):
  - Hospital General de Alicante, Alicante
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Institut Català d'Oncologia - L'Hospitalet, Barcelona
  - Hospital General Castellón, Castelló
  - Hospital Universitario Reina Sofia, Córdoba
  - Complejo Hospitalario de Jaén, Jaén
  - H. U. Insular Gran Canaria, Las Palmas
  - Regional Universitario Carlos Haya, Málaga
  - H Morales Meseguer, Murcia
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Arnau Vilanova Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (7):
  - Kantonsspital Graubünden, Chur
  - HFR Fribourg, Fribourg
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Onkologiezentrum Berner Oberland, Thun
  - Kantonsspital Winterthur, Winterthur
  - Universitätsspital Zürich, Zurich
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Aberdeen
  - Oxford University Hospitals Trust, Oxford
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen LS, Gordon D, Tchekmedyian NS, Yanagihara R, Hirsh V, Krzakowski M, Pawlicki M, De Souza P, Zheng M, Urbanowitz G, Reitsma D, Seaman J. Long-term efficacy and safety of zoledronic acid in the treatment of skeletal metastases in patients with nonsmall cell lung carcinoma and other solid tumors: a randomized, Phase III, double-blind, placebo-controlled trial. Cancer. 2004 Jun 15;100(12):2613-21. doi: 10.1002/cncr.20308. PMID 15197804
- [Background] Tsuya A, Kurata T, Tamura K, Fukuoka M. Skeletal metastases in non-small cell lung cancer: a retrospective study. Lung Cancer. 2007 Aug;57(2):229-32. doi: 10.1016/j.lungcan.2007.03.013. Epub 2007 Apr 23. PMID 17451841
- [Background] Henry DH, Costa L, Goldwasser F, Hirsh V, Hungria V, Prausova J, Scagliotti GV, Sleeboom H, Spencer A, Vadhan-Raj S, von Moos R, Willenbacher W, Woll PJ, Wang J, Jiang Q, Jun S, Dansey R, Yeh H. Randomized, double-blind study of denosumab versus zoledronic acid in the treatment of bone metastases in patients with advanced cancer (excluding breast and prostate cancer) or multiple myeloma. J Clin Oncol. 2011 Mar 20;29(9):1125-32. doi: 10.1200/JCO.2010.31.3304. Epub 2011 Feb 22. PMID 21343556
- [Background] Tan W, Zhang W, Strasner A, Grivennikov S, Cheng JQ, Hoffman RM, Karin M. Tumour-infiltrating regulatory T cells stimulate mammary cancer metastasis through RANKL-RANK signalling. Nature. 2011 Feb 24;470(7335):548-53. doi: 10.1038/nature09707. Epub 2011 Feb 16. PMID 21326202
- [Background] Scagliotti GV, Hirsh V, Siena S, Henry DH, Woll PJ, Manegold C, Solal-Celigny P, Rodriguez G, Krzakowski M, Mehta ND, Lipton L, Garcia-Saenz JA, Pereira JR, Prabhash K, Ciuleanu TE, Kanarev V, Wang H, Balakumaran A, Jacobs I. Overall survival improvement in patients with lung cancer and bone metastases treated with denosumab versus zoledronic acid: subgroup analysis from a randomized phase 3 study. J Thorac Oncol. 2012 Dec;7(12):1823-1829. doi: 10.1097/JTO.0b013e31826aec2b. PMID 23154554
- See also: Sponsor — http://www.etop-eu.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was screened on Jan 12, 2015. On Jan 31, 2018, when accrual to the study was closed, 595 patients were registered in the study by 55 sites in 10 countries. Of the 595 patients who were screened and registered, 514 (86%) were randomized.
Pre-assignment Details: Age ≥ 18 years ECOG performance status 0-2 Histologically or cytologically confirmed advanced stage IV non-small cell lung carcinoma (NSCLC), according to 7th TNM classification Life expectancy of at least 3 months.
Groups:
- None, Standard Chemotherapy Only: 4 - 6 cycles of standard chemotherapy + best supportive care including any bone protective agent except denosumab.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  None, standard chemotherapy only: Possible standard chemotherapies (3 weeks cycles, duration: 4 - 6 cycles):
  Cisplatin 75 mg/m2 as an infusion on day 1 Gemcitabine 1250 mg/m2 as an infusion days 1 and 8 or Carboplatin AUC 5 as an infusion on day 1 Gemcitabine 1000 mg/m2 as an infusion days 1 and 8 or Cisplatin 75 mg/m2 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1 or Carboplatin AUC 5 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1
- Standard Chemotherapy + Denosumab: 4 - 6 cycles of standard chemotherapy + denosumab 120 mg, administered subcutaneously every 3-4 weeks until unacceptable toxicity, patient refusal, or patient's death. Denosumab should be administered on day 1 of each cycle, before or after the administration of chemotherapy. After stop of first-line chemotherapy, denosumab must be continued life-long, regardless of tumour progression and concomitantly with subsequent lines of systemic treatment, as long as tolerable for the patient.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  Denosumab: Denosumab: 120 mg, s.c. every 3-4 weeks (in cycle 1 additional dose on day 8) until unacceptable toxicity, patient refusal or patient's death (max. 4 years 3 months).
Period: Overall Study
Arm/Group | None, Standard Chemotherapy Only | Standard Chemotherapy + Denosumab
Started | 255 | 259
Completed | 252 | 257
Not Completed | 3 | 2
Not completed — Did not start treatment | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | None, Standard Chemotherapy Only | Standard Chemotherapy + Denosumab | Total
Number analyzed (Participants) | 255 | 259 | 514
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 117 | 107 | 224
  >=65 years | 138 | 152 | 290
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 179 | 366
  Male | 68 | 80 | 148
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Histology [Number; unit: participants]
  Squamous | 65 | 70 | 135
  Non-squamous | 187 | 183 | 370
  Mixed | 3 | 6 | 9
Bone metastasis [Number; unit: participants]
  No | 118 | 121 | 239
  Yes | 137 | 138 | 275
ECOG Performance status (PS) [Number; unit: participants] — This tool describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.).
  PS 0: Fully active PS 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  participants
    PS 0/1 (fully active or lightly restricted) | 229 | 230 | 459
    PS 2 (ambulatory and capable of selfcare but unable to carry out work activities) | 26 | 29 | 55
Region [Number; unit: participants]
  Eastern Europe | 18 | 10 | 28
  Western Europe | 153 | 162 | 315
  Southern Europe | 84 | 87 | 171

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: OS will be defined as the time from the date of randomization to the date of death, whatever the cause. The follow-up of participants still alive will be censored at the moment of last follow-up. OS will be reported for all participants in both treatment arms.
Time Frame: Overall survival was measured from the date of randomization to the date of death, whatever the cause, up to a maximum of 56 months
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | None, Standard Chemotherapy Only | Standard Chemotherapy + Denosumab
Number analyzed (Participants) | 255 | 259
years | 0.73 [0.63 to 0.92] | 0.68 [0.62 to 0.87]
Statistical Analysis 1: Comparison: None, Standard Chemotherapy Only vs Standard Chemotherapy + Denosumab; Test type: Superiority — Pre-specified analysis; p = 0.355, Regression, Cox; Cox regression model for treatment effect, analysis adjusted for stratification factors; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.78 to 1.19]

2. Secondary Outcome: Progression-free Survival (PFS) Based on RECIST 1.1
Description: Progression-free survival (PFS) is defined as time from date of randomisation until objective disease progression or death, whichever occurs first. Disease progression and its evaluation are defined based on RECIST 1.1: Progressive disease (PD); > 20% increase in the sum of the longest diameter of target lesions, new lesions or non-equivocal progression in non-target disease.
  If neither event has been observed, then the patient is censored at the date of the last follow up examination.
  Patients with new non-lung cancer malignancy must continue to be followed for progression of the original lung cancer.
  Patients who discontinue treatment prior to documented disease progression, including those who initiate non-protocol therapy prior to progression, will be followed for disease progression and death.
Time Frame: Time from date of randomisation until objective disease progression or death, whichever occurs first, assessed up to a maximum of 56 months
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | None, Standard Chemotherapy Only | Standard Chemotherapy + Denosumab
Number analyzed (Participants) | 255 | 259
years | .39 [.34 to .44] | .39 [.35 to .44]
Statistical Analysis 1: Comparison: None, Standard Chemotherapy Only vs Standard Chemotherapy + Denosumab; Test type: Superiority — Pre-specified analysis; p = 0.459, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.82 to 1.19]

3. Secondary Outcome: Number of Participants With Response (CR+PR) Based on RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  For more details to RECIST 1.1 criteria, see https://recist.eortc.org/
Time Frame: Response of the tumour is defined according to RECIST 1.1 criteria, assessed up to 56 months
Measure: Count of Participants; unit: Participants
Arm/Group | None, Standard Chemotherapy Only | Standard Chemotherapy + Denosumab
Number analyzed (Participants) | 255 | 259
Participants
  Complete response | 1 | 1
  Partial response | 74 | 78
  Stable disease | 101 | 87
  Progressive disease | 51 | 70
  Not evaluable | 27 | 23
  Missing | 1 | 0

4. Secondary Outcome: Toxicity Profile of Denosumab
Description: Number of patients with serious adverse events classified according to NCI CTCAE V4.
Time Frame: Assessed up to 56 months
Measure: Count of Participants; unit: Participants
Arm/Group | None, Standard Chemotherapy Only | Standard Chemotherapy + Denosumab
Number analyzed (Participants) | 255 | 259
Participants
  Patients with serious adverse events | 97 | 138
  Patients without serious adverse events | 158 | 121

5. Secondary Outcome: Overall Survival by Membranous RANK Expression.
Description: Overall survival is defined as time from the date of randomisation until death from any cause. Patients who are still alive at last contact are censored at the date of last follow up.
Time Frame: Up to maximum of 56 months
Population: Information on RANK(L) measurements was available for 463 patients, 229 in chemotherapy alone and 234 in chemotherapy-denosumab arm, among the total 514 patients randomized in the SPLENDOUR trial.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- None, Standard Chemotherapy Only, RANK (+): Membranous RANK(+) patients only, receiving
  4 - 6 cycles of standard chemotherapy + best supportive care including any bone protective agent except denosumab.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  None, standard chemotherapy only: Possible standard chemotherapies (3 weeks cycles, duration: 4 - 6 cycles):
  Cisplatin 75 mg/m2 as an infusion on day 1 Gemcitabine 1250 mg/m2 as an infusion days 1 and 8 or Carboplatin AUC 5 as an infusion on day 1 Gemcitabine 1000 mg/m2 as an infusion days 1 and 8 or Cisplatin 75 mg/m2 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1 or Carboplatin AUC 5 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1
- Standard Chemotherapy + Denosumab, RANK (+): Membranous RANK(+) patients only, receiving
  4 - 6 cycles of standard chemotherapy + denosumab 120 mg, administered subcutaneously every 3-4 weeks until unacceptable toxicity, patient refusal, or patient's death. Denosumab should be administered on day 1 of each cycle, before or after the administration of chemotherapy. After stop of first-line chemotherapy, denosumab must be continued life-long, regardless of tumour progression and concomitantly with subsequent lines of systemic treatment, as long as tolerable for the patient.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  Denosumab: Denosumab: 120 mg, s.c. every 3-4 weeks (in cycle 1 additional dose on day 8) until unacceptable toxicity, patient refusal or patient's death (max. 4 years 3 months).
- None, Standard Chemotherapy Only, RANK (-): Membranous RANK (-) patients only, receiving 4 - 6 cycles of standard chemotherapy + best supportive care including any bone protective agent except denosumab.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  None, standard chemotherapy only: Possible standard chemotherapies (3 weeks cycles, duration: 4 - 6 cycles):
  Cisplatin 75 mg/m2 as an infusion on day 1 Gemcitabine 1250 mg/m2 as an infusion days 1 and 8 or Carboplatin AUC 5 as an infusion on day 1 Gemcitabine 1000 mg/m2 as an infusion days 1 and 8 or Cisplatin 75 mg/m2 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1 or Carboplatin AUC 5 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1
- Standard Chemotherapy + Denosumab, RANK(-): Membranous RANK(-) patients only, receiving
  4 - 6 cycles of standard chemotherapy + denosumab 120 mg, administered subcutaneously every 3-4 weeks until unacceptable toxicity, patient refusal, or patient's death. Denosumab should be administered on day 1 of each cycle, before or after the administration of chemotherapy. After stop of first-line chemotherapy, denosumab must be continued life-long, regardless of tumour progression and concomitantly with subsequent lines of systemic treatment, as long as tolerable for the patient.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  Denosumab: Denosumab: 120 mg, s.c. every 3-4 weeks (in cycle 1 additional dose on day 8) until unacceptable toxicity, patient refusal or patient's death (max. 4 years 3 months).
Arm/Group | None, Standard Chemotherapy Only, RANK (+) | Standard Chemotherapy + Denosumab, RANK (+) | None, Standard Chemotherapy Only, RANK (-) | Standard Chemotherapy + Denosumab, RANK(-)
Number analyzed (Participants) | 77 | 80 | 152 | 154
Months | 7.1 [5.6 to 9.2] | 8.2 [6.6 to 12.5] | 9.1 [6.8 to 11.9] | 7.9 [7.2 to 10.7]

6. Secondary Outcome: Overall Survival by Cytoplasmic RANK Expression.
Description: as for outcome 5
Time Frame: up to a maximum of 56 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- None, Standard Chemotherapy Only, RANK (+): Cytoplasmic RANK(+) patients only, receiving
  4 - 6 cycles of standard chemotherapy + best supportive care including any bone protective agent except denosumab.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  None, standard chemotherapy only: Possible standard chemotherapies (3 weeks cycles, duration: 4 - 6 cycles):
  Cisplatin 75 mg/m2 as an infusion on day 1 Gemcitabine 1250 mg/m2 as an infusion days 1 and 8 or Carboplatin AUC 5 as an infusion on day 1 Gemcitabine 1000 mg/m2 as an infusion days 1 and 8 or Cisplatin 75 mg/m2 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1 or Carboplatin AUC 5 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1
- Standard Chemotherapy + Denosumab, RANK (+): Cytoplasmic RANK(+) patients only receiving
  4 - 6 cycles of standard chemotherapy + denosumab 120 mg, administered subcutaneously every 3-4 weeks until unacceptable toxicity, patient refusal, or patient's death. Denosumab should be administered on day 1 of each cycle, before or after the administration of chemotherapy. After stop of first-line chemotherapy, denosumab must be continued life-long, regardless of tumour progression and concomitantly with subsequent lines of systemic treatment, as long as tolerable for the patient.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  Denosumab: Denosumab: 120 mg, s.c. every 3-4 weeks (in cycle 1 additional dose on day 8) until unacceptable toxicity, patient refusal or patient's death (max. 4 years 3 months).
- None, Standard Chemotherapy Only, RANK (-): Cytoplasmic RANK(-) patients only, receiving
  4 - 6 cycles of standard chemotherapy + best supportive care including any bone protective agent except denosumab.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  None, standard chemotherapy only: Possible standard chemotherapies (3 weeks cycles, duration: 4 - 6 cycles):
  Cisplatin 75 mg/m2 as an infusion on day 1 Gemcitabine 1250 mg/m2 as an infusion days 1 and 8 or Carboplatin AUC 5 as an infusion on day 1 Gemcitabine 1000 mg/m2 as an infusion days 1 and 8 or Cisplatin 75 mg/m2 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1 or Carboplatin AUC 5 as an infusion on day 1 Pemetrexed 500 mg/m2 as an infusion on day 1
- Standard Chemotherapy + Denosumab, RANK (-): Cytoplasmic RANK(-) patients only, receiving
  4 - 6 cycles of standard chemotherapy + denosumab 120 mg, administered subcutaneously every 3-4 weeks until unacceptable toxicity, patient refusal, or patient's death. Denosumab should be administered on day 1 of each cycle, before or after the administration of chemotherapy. After stop of first-line chemotherapy, denosumab must be continued life-long, regardless of tumour progression and concomitantly with subsequent lines of systemic treatment, as long as tolerable for the patient.
  Standard chemotherapy consis of a combination of platinum-based doublet agents plus gemcitabine or pemetrexed.
  Denosumab: Denosumab: 120 mg, s.c. every 3-4 weeks (in cycle 1 additional dose on day 8) until unacceptable toxicity, patient refusal or patient's death (max. 4 years 3 months).
Arm/Group | None, Standard Chemotherapy Only, RANK (+) | Standard Chemotherapy + Denosumab, RANK (+) | None, Standard Chemotherapy Only, RANK (-) | Standard Chemotherapy + Denosumab, RANK (-)
Number analyzed (Participants) | 22 | 19 | 207 | 215
Months | 10.1 [6.7 to 20.7] | 8.5 [3.5 to 18.6] | 7.8 [6.2 to 10.4] | 7.9 [7.1 to 10.1]

ADVERSE EVENTS:
Time Frame: On day 1 of every 3-week treatment cycle, at the end of treatment, every 6-8 weeks thereafter until end of study, for a maximum of 56 months.
Arm/Group | None, Standard Chemotherapy Only | Standard Chemotherapy + Denosumab
All-Cause Mortality (participants affected / at risk) | 178/255 | 177/259
Serious Adverse Events (participants affected / at risk) | 97/255 | 138/259
Other Adverse Events (participants affected / at risk) | 235/255 | 246/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | None, Standard Chemotherapy Only (N=255) | Standard Chemotherapy + Denosumab (N=259)
ANAEMIA (Blood and lymphatic system disorders) | 14 (16) | 9 (11)
ANAEMIA OF MALIGNANT DISEASE (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 10 (11)
HAEMATOTOXICITY (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 9 (10) | 8 (8)
NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 5 (5) | 10 (12)
SPLENIC HAEMORRHAGE (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 9 (10) | 13 (14)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 2 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 2 (2)
APLASIA (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 3 (3)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 4 (4)
DIARRHOEA (Gastrointestinal disorders) | 7 (7) | 8 (8)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 2 (2)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GINGIVAL DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
IMMUNE-MEDIATED ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 6 (8) | 15 (19)
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (4) | 11 (16)
ASTHENIA (General disorders) | 3 (3) | 3 (3)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
CONDITION AGGRAVATED (General disorders) | 0 (0) | 1 (1)
DEATH (General disorders) | 0 (0) | 5 (5)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0)
EUTHANASIA (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 6 (6) | 4 (5)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 5 (5) | 6 (7)
HYPERTHERMIA (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 3 (3) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 3 (3) | 7 (7)
PYREXIA (General disorders) | 5 (5) | 2 (2)
SUDDEN DEATH (General disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (3) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1)
BACTERIAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 0 (0)
DEVICE OCCLUSION (Infections and infestations) | 1 (1) | 1 (1)
ENTEROBACTER INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FUNGAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
HERPES SIMPLEX OESOPHAGITIS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 2 (2)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2)
NECROTISING FASCIITIS (Infections and infestations) | 1 (1) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 2 (2)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 2 (2) | 0 (0)
PAROTITIS (Infections and infestations) | 0 (0) | 1 (1)
PICORNAVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 9 (9) | 17 (17)
PNEUMONIA NECROTISING (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (9) | 4 (4)
SEPSIS (Infections and infestations) | 4 (4) | 6 (7)
SEPTIC SHOCK (Infections and infestations) | 3 (3) | 5 (5)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
TRACHEOBRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5) | 2 (2)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
OXYGEN SATURATION DECREASED (Investigations) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 7 (7)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ENDOCRINE NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LYMPHANGIOSIS CARCINOMATOSA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR ASSOCIATED FEVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (3)
DIZZINESS (Nervous system disorders) | 2 (2) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGICAL DECOMPENSATION (Nervous system disorders) | 0 (0) | 1 (1)
PERONEAL NERVE PALSY (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 3 (3)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
DEVICE BREAKAGE (Product Issues) | 0 (0) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 2 (2)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 4 (4) | 4 (4)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 6 (7) | 4 (4)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OESOPHAGOBRONCHIAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)
ISCHAEMIA (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | None, Standard Chemotherapy Only (N=255) | Standard Chemotherapy + Denosumab (N=259)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 13 (17)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 (2) | 0 (0)
ASYSTOLE (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 4 (4) | 6 (7)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 3 (4)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC TOXICITY (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1) | 1 (1)
CIRCULATORY INSUFFICIENCY (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY INSUFFICIENCY (Cardiac disorders) | 0 (0) | 1 (1)
EXTRASYSTOLEN (Cardiac disorders) | 0 (0) | 1 (1)
HEART FAILURE (Cardiac disorders) | 1 (1) | 2 (3)
MOBITZ (TYPE) II ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 2 (2)
PERICARDIAL TAMPONADE (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 3 (3) | 3 (3)
SUPRAVENTRICULAR EXTRASYSTOLE (Cardiac disorders) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (1)
VALVULAR HEART DEFECT (Cardiac disorders) | 1 (1) | 0 (0)
DISORDERS OF EQUILIBRUM (Ear and labyrinth disorders) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1)
EXTERNAL EAR INFLAMMATION (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING IMPAIRED (Ear and labyrinth disorders) | 6 (6) | 3 (3)
TINNITUS (Ear and labyrinth disorders) | 6 (9) | 3 (5)
VERTIGO (Ear and labyrinth disorders) | 8 (9) | 13 (20)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 1 (1)
CUSHINGOID (Endocrine disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 3 (3)
THYROIDITIS (Endocrine disorders) | 0 (0) | 1 (1)
BAD VISION RIGHT EYE (Eye disorders) | 1 (1) | 0 (0)
BLURRED VISION (Eye disorders) | 3 (3) | 6 (6)
CONJUCTIVITIS (Eye disorders) | 1 (1) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 7 (8) | 6 (9)
DRY EYE (Eye disorders) | 4 (4) | 6 (6)
EXTRAOCULAR MUSCLE PARESIS (Eye disorders) | 1 (1) | 0 (0)
EYE DISORDER OTHER- HEMORRHAGE EYE (Eye disorders) | 0 (0) | 1 (1)
EYE IRRITATION (Eye disorders) | 1 (1) | 0 (0)
EYE PAIN (Eye disorders) | 2 (2) | 3 (3)
INFLAMMATION RIGHT EYE (Eye disorders) | 0 (0) | 1 (1)
INTENSIFIED TEAR FLUID (Eye disorders) | 1 (1) | 0 (0)
OSCILLOPSIA (Eye disorders) | 0 (0) | 1 (1)
PAPILLEDEMA (Eye disorders) | 0 (0) | 1 (1)
REDUCED VISION (Eye disorders) | 0 (0) | 1 (1)
SUB CONJUNCTIVAL HEMORRHAGE(LEFT EYE) (Eye disorders) | 1 (1) | 0 (0)
SUBCONJUNCTIVAL HEMORRHAGE RIGHT EYE (Eye disorders) | 0 (0) | 1 (1)
VISUAL DISTURBANCES (Eye disorders) | 1 (1) | 0 (0)
WATERING EYES (Eye disorders) | 8 (11) | 7 (10)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 14 (16) | 21 (35)
ANAL ABSCESS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ANAL FISTULA (Gastrointestinal disorders) | 0 (0) | 2 (2)
ANAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1)
ANAL MUCOSITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLEEDING SPLEEN (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLOATING (Gastrointestinal disorders) | 1 (1) | 1 (2)
CHEILITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 3 (3) | 3 (3)
COLONDIVERTICULOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 54 (71) | 69 (94)
CONTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 41 (57) | 53 (74)
DIGESTION PROBLEMS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIVERTICULITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIVERTICULOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 5 (5)
DYSGEUSIA (Gastrointestinal disorders) | 1 (2) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 7 (10) | 7 (8)
DYSPHAGIA (Gastrointestinal disorders) | 9 (12) | 9 (10)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 2 (4)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1)
ESOPHAGEAL FISTULA (Gastrointestinal disorders) | 1 (1) | 1 (1)
ESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ESOPHAGEAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
ESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ESOPHAGITIS (Gastrointestinal disorders) | 3 (6) | 2 (2)
FATIGUE (Gastrointestinal disorders) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 3 (3) | 3 (4)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 (4) | 9 (10)
GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL DISORDERS -OTHER:UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 4 (5) | 4 (4)
ILEUS (Gastrointestinal disorders) | 2 (2) | 0 (0)
MUCOSITIS ORAL (Gastrointestinal disorders) | 34 (38) | 42 (62)
NAUSEA (Gastrointestinal disorders) | 91 (147) | 92 (162)
NEUTROPENIC ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 4 (4)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 0 (0) | 4 (4)
PERIOTONDAL DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 0 (0)
RECTAL MUCOSITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
SIGMADIVERTICULITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
SORE, SWOLLEN TONGUE (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 10 (10) | 2 (2)
TOOTH EXTRACTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 2 (2)
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (2)
VOMITING (Gastrointestinal disorders) | 45 (61) | 45 (67)
VOMITTING (Gastrointestinal disorders) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (General disorders) | 1 (1) | 0 (0)
ALTERATION OF GENERAL CONDITION (General disorders) | 1 (2) | 0 (0)
ALTERATION OF GENERAL STATUS (General disorders) | 0 (0) | 1 (1)
BACK PAIN (General disorders) | 1 (1) | 0 (0)
BONE PAIN (General disorders) | 0 (0) | 1 (1)
CHEST WALL PAIN (General disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 5 (6)
CONSTITUTIONAL SYNDROME (General disorders) | 1 (2) | 0 (0)
CRAMPS (General disorders) | 1 (1) | 0 (0)
DEATH NOS (General disorders) | 0 (0) | 1 (1)
DECLINE IN GENERAL HEALTH STATUS (General disorders) | 0 (0) | 1 (1)
DECLINE IN HEALTH STATUS (General disorders) | 0 (0) | 1 (1)
DECREASED MOBILITY (General disorders) | 0 (0) | 1 (1)
DETERIORATION IN HEALTH (General disorders) | 1 (1) | 0 (0)
DETERIORATION OF GENERAL STATE (General disorders) | 0 (0) | 1 (1)
DRY MUCOSAE (General disorders) | 1 (1) | 0 (0)
DRY MUCOUS MEMBRANES (General disorders) | 0 (0) | 1 (1)
EDEMA FACE (General disorders) | 1 (1) | 2 (2)
EDEMA LIMBS (General disorders) | 31 (43) | 27 (37)
FACIAL PAIN (General disorders) | 0 (0) | 3 (3)
FATIGUE (General disorders) | 120 (214) | 133 (287)
FEVER (General disorders) | 22 (23) | 21 (30)
FLU LIKE SYMPTOMS (General disorders) | 7 (9) | 5 (6)
GAIT DISTURBANCE (General disorders) | 2 (2) | 1 (1)
GENERAL DETERIORATION (General disorders) | 2 (3) | 2 (3)
GENERAL DISORDERS + ADMINISTRATION SITE CONDITIONS (General disorders) | 1 (2) | 1 (1)
GENERAL HEALTH DETERIORATION (General disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1)
GENERALIZED EDEMA (General disorders) | 0 (0) | 1 (1)
HEADACHE (General disorders) | 0 (0) | 1 (1)
HEALTH DETERIORATION (General disorders) | 1 (1) | 0 (0)
HOT FLASHES DURING THE NIGHT (General disorders) | 1 (1) | 0 (0)
INFUSION SITE EXTRAVASATION (General disorders) | 1 (1) | 0 (0)
INJECTION SITE REACTION (General disorders) | 2 (2) | 1 (1)
IRRITABILITY (General disorders) | 1 (1) | 0 (0)
LOCALIZED EDEMA (General disorders) | 3 (3) | 5 (6)
LOSS OF APPETITE (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 12 (16) | 19 (23)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 1 (1)
NIGHT SWEATS (General disorders) | 3 (3) | 1 (1)
NON CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 15 (18) | 21 (24)
PAIN (General disorders) | 33 (50) | 33 (55)
PAIN IN EXTREMITY (General disorders) | 1 (1) | 2 (2)
PAIN OTHER - LEFT GROIN (General disorders) | 1 (1) | 0 (0)
PROGRESSION OF DISEASE (General disorders) | 1 (2) | 0 (0)
SUBFEBRILE TEMPERATURES (General disorders) | 1 (1) | 0 (0)
SUDDEN DEATH NOS (General disorders) | 0 (0) | 1 (1)
SWEAT (General disorders) | 0 (0) | 1 (1)
SWOLLEN FACE (General disorders) | 0 (0) | 1 (1)
WORSENING OF CLINICAL CONDITION (General disorders) | 0 (0) | 1 (1)
WORSENING OF GENERAL CONDITION (General disorders) | 1 (1) | 2 (2)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (3) | 0 (0)
HEPATIC PAIN (Hepatobiliary disorders) | 0 (0) | 1 (1)
LIVER CONGESTION (Hepatobiliary disorders) | 1 (1) | 0 (0)
LIVER LIPOMAS (Hepatobiliary disorders) | 1 (1) | 0 (0)
TRANSAMINITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
WORSENING LIVER FUNCTION (Hepatobiliary disorders) | 0 (0) | 1 (1)
ALLERGIC REACTION (Immune system disorders) | 5 (5) | 5 (5)
INTOLERANCE OF RED BLOOD CELL CONCENTRATE (Immune system disorders) | 0 (0) | 1 (1)
RIGHT CERVICAL LYMPHADENOPATHY (Immune system disorders) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1)
BLADDER INFECTION (Infections and infestations) | 1 (1) | 1 (1)
BRONCHIAL INFECTION (Infections and infestations) | 9 (12) | 11 (14)
CATHETER RELATED INFECTION (Infections and infestations) | 1 (1) | 1 (1)
ENTEROBACTER CLOACAO INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 1 (1)
ESOPHAGEAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FLU LIKE SYMPTOMS (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 3 (3)
INFECTION OF UNCLEAR GENESIS (Infections and infestations) | 1 (1) | 0 (0)
INFECTIONS & INFESTATIONS OTHER - HEAD COLD (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA A (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA B (Infections and infestations) | 1 (1) | 0 (0)
JOINT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
LIP INFECTION (Infections and infestations) | 4 (4) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 24 (34) | 40 (55)
MENINGITIS (Infections and infestations) | 1 (1) | 0 (0)
MUCOSAL INFECTION (Infections and infestations) | 1 (1) | 4 (5)
MYCOSIS (IN OESOPHAGUS) (Infections and infestations) | 1 (1) | 0 (0)
ORAL VIRAL EVENT (Infections and infestations) | 1 (1) | 0 (0)
PAPULOPUSTULAR RASH (Infections and infestations) | 0 (0) | 1 (1)
PAROTIDITIS (Infections and infestations) | 1 (1) | 0 (0)
PENILE INFECTION (Infections and infestations) | 1 (1) | 1 (1)
PERSISTING INFLAMMATION DUE TO MALIGNANCY (Infections and infestations) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 2 (2) | 3 (3)
PHLEBITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1)
PLEURAL INFECTION (Infections and infestations) | 2 (2) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 1 (1) | 3 (3)
RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
RHINITIS INFECTIVE (Infections and infestations) | 3 (3) | 2 (2)
SCROTAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 10 (15) | 11 (16)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 2 (2) | 1 (1)
SKIN INFECTION (Infections and infestations) | 3 (4) | 7 (9)
STOMA SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STOMATITIS (Infections and infestations) | 0 (0) | 1 (1)
SUSPECTED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SUSPECTED INFECTION OF RICKHAM RESERVOIR (Infections and infestations) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (2)
TRACHEITIS (Infections and infestations) | 1 (1) | 1 (1)
UNCLEAR INFECT-FOCUS, NO GERM-EVIDENCE (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 18 (22) | 24 (33)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URETHRAL INFECTION (Infections and infestations) | 0 (0) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 9 (9) | 11 (12)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VULVAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 2 (2)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ARTIPHICIAL SPHINTER RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DERMATITIS RADIATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
FRACTURE (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
HIP DISLOCATION (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
OCCLUSION OF STENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POSTTHORACOTOMY SYNDROM (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WOUND HAND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (5) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) | 4 (4)
C REACTIVE PROTEIN (Investigations) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 2 (2) | 2 (2)
CARBON MONOXIDE DIFFUSING CAPACITY DECREASED (Investigations) | 0 (0) | 1 (1)
CREATININE INCREASED (Investigations) | 1 (1) | 1 (1)
ELEVATED C REACTIVE PROTEIN VALUES (Investigations) | 1 (1) | 0 (0)
EOSINOPHIL COUNT INCREASED (Investigations) | 0 (0) | 1 (1)
GGT INCREASED (Investigations) | 7 (9) | 3 (6)
HYPOMAGNESEMIA (Investigations) | 1 (1) | 0 (0)
IRON DEFICIENCY (Investigations) | 0 (0) | 1 (1)
LDH INCREASED (Investigations) | 0 (0) | 1 (1)
LEUCOCYTES AND C REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 1 (1)
LOSS OF WEIGHT (Investigations) | 1 (1) | 0 (0)
LOW VITAMIN D (Investigations) | 0 (0) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 1 (3)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
RAISED CRP (Investigations) | 0 (0) | 1 (1)
URAEMIA (Investigations) | 0 (0) | 1 (1)
WEIGHT LOSS (Investigations) | 0 (0) | 1 (1)
WEIGHT GAIN (Investigations) | 34 (56) | 50 (97)
WEIGHT LOSS (Investigations) | 71 (97) | 95 (172)
ANOREXIA (Metabolism and nutrition disorders) | 61 (84) | 68 (104)
APPETITE INCREASED (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
CACHEXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (4) | 9 (11)
DIABETIC KETOSIS WITH METABOLIC ALKALOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ELECTROLYTE DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
EXSICCOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
GLUCOSE INTOLERANCE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERCHOLESTEROLEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 5 (6) | 5 (19)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
HYPERURICEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 7 (9) | 11 (15)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 9 (23) | 7 (11)
HYPONATREMIA (Metabolism and nutrition disorders) | 8 (9) | 9 (15)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 3 (3) | 10 (19)
LOSS OF APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
PSEUDOGOUT (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (6) | 11 (13)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 22 (33) | 24 (33)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 18 (21) | 12 (18)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (10)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
HERNIATED DISC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
LEFT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
MUSCLE WEAKNESS UPPER LIMB (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN - RIGHT HIP (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 12 (14) | 14 (16)
PAIN LEFT AXILLA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN OTHER - RIGHT GLUTEAL AREA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN RIGHT MANDIBULA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ADENOPATHY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BRAIN METASTASES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SEEPING METASTASIS UNDER SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TENDERNESS AT SITE OF LUNG MASS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 7 (7)
AKATHISIA (Nervous system disorders) | 1 (1) | 1 (1)
AMNESIA (Nervous system disorders) | 1 (1) | 0 (0)
APHONIA (Nervous system disorders) | 3 (3) | 1 (1)
ATAXIA (Nervous system disorders) | 0 (0) | 6 (7)
CEREBROSPINAL FLUID FISTULA (Nervous system disorders) | 1 (1) | 0 (0)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1) | 0 (0)
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 12 (12) | 10 (11)
DYSDIADOCHOKINESIS (Nervous system disorders) | 0 (0) | 1 (1)
DYSESTHESIA (Nervous system disorders) | 2 (2) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 27 (28) | 23 (41)
DYSPHASIA (Nervous system disorders) | 1 (1) | 2 (2)
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 1 (1) | 1 (1)
FACIAL NERVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 15 (19) | 19 (20)
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 0 (0) | 2 (3)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (6)
MOVEMENTS INVOLUNTARY (Nervous system disorders) | 1 (1) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 2 (2)
NUMBNESS ON THE TIP OF FINGERS (Nervous system disorders) | 0 (0) | 1 (1)
OCULOMOTOR NERVE DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
PARESTHESIA (Nervous system disorders) | 9 (10) | 9 (9)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 3 (5) | 3 (7)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 11 (11) | 14 (18)
POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 2 (2) | 0 (0)
RIGHT SIDED SCIATICA (Nervous system disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 2 (3)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 3 (3)
STROKE (Nervous system disorders) | 1 (1) | 3 (6)
SYNCOPE (Nervous system disorders) | 5 (5) | 4 (5)
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 1 (1) | 1 (1)
TREMOR (Nervous system disorders) | 2 (2) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 2 (2)
ANXIETY (Psychiatric disorders) | 9 (13) | 8 (10)
CONFUSION (Psychiatric disorders) | 4 (4) | 8 (9)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 5 (7) | 7 (8)
HALLUCINATIONS (Psychiatric disorders) | 2 (2) | 0 (0)
INSOMNIA (Psychiatric disorders) | 12 (15) | 12 (14)
PSYCHIATRIC DISORDER OTHER: ADAPTIVE DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 8 (11) | 4 (5)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 2 (2) | 3 (4)
CYSTITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 1 (1) | 1 (1)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 1 (1) | 2 (2)
NYCTURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL AND URINARY DISORDERS - RENAL PAIN (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL INSUFFICIENCY (Renal and urinary disorders) | 2 (3) | 1 (1)
URINARY FREQUENCY (Renal and urinary disorders) | 0 (0) | 2 (2)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 2 (2)
URINARY RETENTION (Renal and urinary disorders) | 2 (2) | 1 (1)
URINARY TRACT INFECTION (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 2 (3) | 0 (0)
URINARY TRACT PAIN (Renal and urinary disorders) | 3 (3) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
DYSMENORRHEA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 2 (2)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PENILE PAIN (Reproductive system and breast disorders) | 2 (2) | 0 (0)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ADULT RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (6)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
BRONCHIAL STRICTURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRONCHOPULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
BRONCHOPULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 13 (18)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 33 (43) | 56 (81)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 62 (80) | 72 (108)
EMPHYSEMA LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 11 (11)
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
LARYNGEAL HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
LARYNGEAL MUCOSITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LUNG INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ORTHOPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PAIN LARYNX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PHARYNGEAL MUCOSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (14)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (10)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 7 (8)
RHINITIS SICCA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RIGHT BASAL HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RIGHT PULMONARY HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RUNNING NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
WHEEZE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
ACTINITIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 (6) | 9 (10)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CELLULITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DARK SKIN DISCOLORATION AXILLAR, SHOULDER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7)
ECZEMA ARMS AND ABDOMINAL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ERYSIPELAS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 4 (4) | 8 (8)
EXANTHEMA BOTH ARMS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
FACIAL WOUND (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
FRAGILITY ON NAILS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HAIR WEAKNESS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (6)
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PERIANAL IRRITATION,WARTS BACK /ONE WART RIGHT EYE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PERIORBITAL EDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 7 (12) | 7 (7)
PSORIASIS REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (10)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 8 (10) | 14 (17)
RASH ON ARMS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3)
TICK BITE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
PAIN STENT (Surgical and medical procedures) | 1 (1) | 0 (0)
PLEURX (Surgical and medical procedures) | 0 (0) | 1 (1)
TOOTH EXTRACTION (Surgical and medical procedures) | 0 (0) | 1 (1)
ARTERIAL HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
HEMATOMA (Vascular disorders) | 2 (3) | 3 (4)
HOT FLASHES (Vascular disorders) | 2 (2) | 6 (6)
HOT FLASHES - RIGHT ARM (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 96 (218) | 109 (326)
HYPERTENTION (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 6 (6) | 9 (10)
LYMPH LEAKAGE (Vascular disorders) | 0 (0) | 1 (1)
LYMPHEDEMA (Vascular disorders) | 0 (0) | 1 (2)
PERIPHERAL ISCHEMIA (Vascular disorders) | 2 (5) | 0 (0)
PHLEBITIS (Vascular disorders) | 3 (4) | 2 (2)
RAYNAUD (Vascular disorders) | 0 (0) | 1 (1)
RAYNAUD'S DISEASE (Vascular disorders) | 1 (1) | 0 (0)
RENAL INFARCTION (Vascular disorders) | 0 (0) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 13 (15) | 14 (16)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 1 (1) | 0 (0)
VASCULAR SCLEROSIS (Vascular disorders) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study steering committee decided to close the study prematurely due to poor accrual. The primary analysis is therefore underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPLENDOUR Steering Committee will be responsible for review and approval of any publication of results from this trial.

The SPLENDOUR Steering Committee will decide the appropriate journal and corresponding author(s).

The SPLENDOUR Steering Committee will decide on authorship of the manuscript. No other participating group or institution should publish its own data on therapy results prior to the major publication.

DOCUMENTS (2):
  • Study Protocol (2014-04-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT02129699/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT02129699/SAP_001.pdf